CLINICAL TRIAL: NCT01988064
Title: Comparison of the Short-term Efficacy of Two Training Methods (Face to Face vs. Group Training) on Pulse Rate Taking in Patients With Cardiovascular Diseases, a Randomized Trial.
Brief Title: Face to Face vs. Group Training Methods on Pulse Rate Taking in Patients With Cardiovascular Diseases.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Saeed Alipour Parsa, Alipour Parsa S., Assistant professor of cardiology, Cardiovascular Research Center, Modarres hospital, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: sbcvrc-106-1014
Record Dates: First submitted 2013-11-04; First posted 2013-11-20 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Arrythmia
Keywords: pulse rate; patient education; training
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Sensitivity Training Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Face-to-face training (Experimental): One-to-one face-to-face training on calculating the pulse rate and detecting pulse abnormalities performed by the nurse.
  Interventions: Other: Face-to-face training
- Group training (Experimental): Group training using a tutorial film on calculating the pulse rate and detecting pulse abnormalities.
  Interventions: Other: Group training

INTERVENTIONS:
Other: Face-to-face training — One-to-one face-to-face training on calculating the pulse rate and detecting abnormalities.
  Arms: Face-to-face training
Other: Group training — Group training using a tutorial film on calculating the pulse rate and detecting abnormalities.
  Arms: Group training

SUMMARY:
The aim of this study is to compare the efficacy of group training using a tutorial film and one-to-one face-to-face training in calculating the pulse rate and detecting irregularity in the pulse rhythm in patients with cardiovascular diseases.

DETAILED DESCRIPTION:
Pulse rate self-examination can provide a fairly good assessment of the patient's condition and helps the physician with drug dosage adjustment in patients with cardiac problems.

This study will be conducted in the Cardiology wards of Modarres and Loghman hospitals in Tehran. These are two educational general referral hospitals of Shahid Beheshti University of medical sciences covering northern and southern part of Tehran, the capital of Iran respectively.

After obtaining a written consent the patients will randomly assign into two groups using random number table. One group will receive a 20-minute face-to-face training session by a nurse on how to calculate the pulse rate in a minute and detect irregularities in the pulse rhythm whereas a 10-minute tutorial film with the same content will be shown to the other group.

Three practical test sessions are arranged for each patient, before the training session, right after the training session and at least 48 hours after the training session. The tests contain two parts and evaluate the patients' ability in calculating the exact pulse rate in a minute and detecting irregularities in the pulse rhythm.

A special data-collecting questionnaire is designed for this study. This questionnaire contains background information such as sex, age, and literacy level as well as the practical test results. Data gathering process will be performed by nurses in these hospitals. Nurses, who participate in this study, will attend in briefing sessions on how to fill the data-collecting questionnaires.

The sample size consists of 300 patients who admitted in Cardiology ward (200 in Modarres hospital and 100 in Loghman hospital). The data will be inserted to the computer and the variables will be compared within and between groups using SPSS software version 16.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in cardiology ward
* Literacy (ability to read and write)

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-04 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Ability to calculated the pulse rate correctly and detected pulse irregularity | The outcome will be measured on three distinct time points; before the training session(base line), right after the training session, and at least 48 hours after the training session
  The number of participants who can calculate the pulse rate correctly and detect pulse irregularity, and the participants' improvement in the ability to calculated the pulse rate correctly and detected pulse irregularity on the three time points, will be compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Habibolah Saadat, Professor of cardiology, Principal Investigator — Cardiovascular research center, Modarres hospital, Shahid Beheshti University of Medical Sciences
Locations (1):
- Cardiovascular research center, Modarres hospital., Tehran, Tehran Province, Iran

REFERENCES:
- [Background] Munschauer FE 3rd, Sohocki D, Smith Carrow S, Priore RL. A community education program on atrial fibrillation: implications of pulse self-examination on awareness and behavior. J Stroke Cerebrovasc Dis. 2004 Sep-Oct;13(5):208-13. doi: 10.1016/j.jstrokecerebrovasdis.2004.08.001. PMID 17903977
- [Background] Hwu YJ, Coates VE, Lin FY. A study of the effectiveness of different measuring times and counting methods of human radial pulse rates. J Clin Nurs. 2000 Jan;9(1):146-52. doi: 10.1046/j.1365-2702.2000.00350.x. PMID 11022503
- [Background] Breckwoldt J, Schloesser S, Arntz HR. Perceptions of collapse and assessment of cardiac arrest by bystanders of out-of-hospital cardiac arrest (OOHCA). Resuscitation. 2009 Oct;80(10):1108-13. doi: 10.1016/j.resuscitation.2009.06.028. Epub 2009 Jul 25. PMID 19632755